CLINICAL TRIAL: NCT01163630
Title: A Phase I, Open-label, Randomized, Single-center, 2-way Crossover Food Interaction Study To Assess the Effect of Food on the Pharmacokinetics of the Fixed Dose Combination Capsule of Esomeprazole 20 mg/Acetylsalicylic Acid 81 mg
Brief Title: Food Interaction Study To Assess the Effect of Food on the Pharmacokinetics of Esomeprazole 20 mg/Acetylsalicylic Acid 81 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D961FC00009
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Effect of Food; Pharmacokinetics
Keywords: open label, randomized; single-center; 2-way crossover; food interaction study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): esomeprazole 20mg/ASA 81 mg FDC after a 10-hour fast
  Interventions: Drug: esomeprazole/ASA Fixed Dose Combination (FDC)
- 2 (Experimental): esomeprazole 20mg/ASA 81 mg FDC 30 minutes after start of a high-fat, high-calorie breakfast
  Interventions: Drug: esomeprazole/ASA Fixed Dose Combination (FDC)

INTERVENTIONS:
Drug: esomeprazole/ASA Fixed Dose Combination (FDC) — esomeprazole 20 mg/ASA 81 mg oral capsule

SUMMARY:
The purpose of the study is to investigate the effects of food, in comparison to fasting conditions, on the extent and rate of absorption of acetylsalicylic acid (ASA) and esomeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who provide informed consent prior to any study-related procedures. Females must be of non-child bearing potential.
* Weight of 50-95kg, inclusive, and a BMI between 19-30 kg/m2, inclusive.
* No clinically significant abnormal findings as judged by the Investigator on enrollment physical exam.

Exclusion Criteria:

* Recent history of any clinically significant illness as judged by the Investigator within two weeks prior to enrolling in the study
* History of heart, kidney, liver. or gastrointestinal disease considered to be significant as judged by the Investigator
* Moderate to heavy smoking or other nicotine use (greater than 10 cigarettes per day or corresponding amount of nicotine)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of food on the extent and rate of absorption of ASA and esomeprazole after a single dose administration of esomeprazole 20mg/ASA 81 mg FDC in healthy volunteers by assessment of AUC, AUC(0-t), and Cmax | Blood samples for ASA and SA analyses will be taken at predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 5, 6, 8, 10, 12, and 14 hours after dose administration
To investigate the effects of food on the extent and rate of absorption of ASA and esomeprazole after a single dose administration of esomeprazole 20mg/ASA 81 mg FDC in healthy volunteers by assessment of AUC, AUC(0-t), and Cmax | Blood samples for esomeprazole analysis will be taken at predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11, 12, 13, and 14 hours after dose adminstration

SECONDARY OUTCOMES:
To investigate PK of ASA and esomeprazole by assessment of tmax and t1/2λz under fed and fasting conditions. | Blood samples for ASA and SA analyses will be taken at predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 5, 6, 8, 10, 12, and 14 hours after dose administration
To investigate the PK of ASA metabolite salicylic acid (SA) by assessment of AUC, AUC(0-t), Cmax, tmax and t1/2λz under fed and fasting conditions. | Blood samples for ASA and SA analyses will be taken at predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 5, 6, 8, 10, 12, and 14 hours after dose administration
To assess the safety and tolerability of esomeprazole 20mg/ASA 81 mg FDC. | AEs will be collected from the time of randomization up to and including the follow-up visit. SAEs will be recorded from the time of informed consent up to and including the follow up visit
To investigate the PK of ASA metabolite salicylic acid (SA) by assessment of AUC, AUC(0-t), Cmax, tmax and t1/2λz under fed and fasting conditions. | Blood samples for esomeprazole analysis will be taken at predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 9, 10, 11, 12, 13, and 14 hours after dose adminstrationy.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Craven, MD, Principal Investigator — Quintiles, Inc.; Ken Price, Study Director — AstraZeneca; Mirjana Kujacic, Study Director — AstraZeneca
Locations (1):
- Research Site, Oveland Park, Kansas, United States